CLINICAL TRIAL: NCT04695665
Title: The Effectiveness of McGill's Method in the Treatment of Vertebrogenic Algic Syndrome
Brief Title: Therapy of Pain Syndromes According to McGill's Method in Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Malá Jitka, assistant professor, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vlasák, McGill
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Vertebrogenic Pain Syndrome
Keywords: pain syndrome; efficiency; stabilization; McGill method
MeSH Terms: conditions — Back Pain; Somatoform Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cervical pain (Active Comparator): Only patients with positive Cervical pain syndrome.
  Interventions: Other: Cervical pain
- Thoracic pain (Active Comparator): Only patients with positive Thoracic pain syndrome.
  Interventions: Other: Thoracic pain
- Lumbar pain (Active Comparator): Only patients with positive Lumbar pain syndrome.
  Interventions: Other: Lumbar pain

INTERVENTIONS:
Other: Cervical pain — Exercise program for cervical spine according to McGill's approach.
  Arms: Cervical pain
Other: Thoracic pain — Exercise program for thoracic spine according to McGill's approach.
  Arms: Thoracic pain
Other: Lumbar pain — Exercise program for lumbar spine according to McGill's approach.
  Arms: Lumbar pain

SUMMARY:
The goal of this study is to determine the applicability of McGill ́s method to patients with diagnoses, collectively referred to as Vertebrogenic Algic syndrome, by comparing the measured data of proband with different diagnosis locations Vertebrogenic Algic syndrome in the Czech Republic.

DETAILED DESCRIPTION:
This is a pilot experimental research involving 10 probands diagnosed with Vertebrogenic Algic syndrome in the cervical spine, 10 probands diagnosed with Vertebrogenic Algic syndrome in the thoracic spine and 10 probands diagnosed with Vertebrogenic Algic syndrome in the lumbar spine. Each participant undergo a kinesiological examination according to the McGill ́s principles together with an SF-36 questionnaire. Measured values are compared and provided a basis for testing the hypotheses. The study uses methods of research, observation, querying and comparison of collected data.

ELIGIBILITY:
Inclusion Criteria:

* cervical pain syndrome
* thoracic pain syndrome
* lumbar pain syndrome

Exclusion Criteria:

* red falgs

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Pain relief | 4 weeks, 2 times a week exercising for 60 minutes
  change in pain perception measured on a visual analog scale - from 0 (without pain) to 10 (maximum pain)
multi-segmental efficiency | 4 weeks
  comparison of the effectiveness of therapy of the three evaluated groups against each other by Short Form (SF36) Healthy survey questionnaire, the scale from 100 to 900, lower value indicate a higher effect

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, Ph.D., Principal Investigator — Charles University, Faculty of physical education and sport
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No